CLINICAL TRIAL: NCT03334617
Title: An Open-Label, Multi-Drug, Biomarker-Directed, Multi-Centre Phase II Umbrella Study in Patients With Non-Small Cell Lung Cancer, Who Progressed on an Anti-PD-1/PD-L1 Containing Therapy (HUDSON).
Brief Title: Phase II Umbrella Study of Novel Anti-cancer Agents in Participants With NSCLC Who Progressed on an Anti-PD-1/PD-L1 Containing Therapy
Acronym: HUDSON
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6185C00001; 138050 (Registry Identifier: IND); 2023-509004-15-00 (Other: EU CT number); 2017-002208-28 (EudraCT Number)
Record Dates: First submitted 2017-09-22; First posted 2017-11-07 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-small cell lung cancer; NSCLC; anti-PD-1/PD-L1; umbrella study; Durvalumab; MEDI4736; Olaparib; AZD2281; AZD9150; AZD6738; Vistusertib; AZD2014; Oleclumab; MEDI9447; Trastuzumab deruxtecan; DS-8201a; cediranib; AZD2171
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; danvatirsen; ceralasertib; vistusertib; olaparib; trastuzumab deruxtecan; cediranib

STUDY DESIGN:
Intervention Model Description: This is an open-label, multi-centre, umbrella Phase II study in participants with metastatic NSCLC who have progressed on an anti-PD-1/PD-L1 containing therapy. This study is modular in design, allowing initial assessment of the efficacy, safety, and tolerability of multiple treatment arms.
  Within each module, there will be treatment cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (22):
- Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg (Experimental): Participants with detectable aberrations, mutation detected in a homologous recombination repair gene (HRRm) will receive IV infusion of durvalumab 1500 mg every 4 weeks (Q4W) in combination with oral olaparib 300 mg (2 × 150 mg) tablets twice a day (BD) until disease progression is confirmed.
  Interventions: Drug: Durvalumab; Drug: Olaparib
- Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg (Experimental): Participants with detectable aberrations in liver kinase B1 (LKB1) will receive IV infusion of durvalumab 1500 mg Q4W in combination with oral olaparib 300 mg (2 × 150 mg) tablets BD until disease progression is confirmed.
  Interventions: Drug: Durvalumab; Drug: Olaparib
- Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg (Experimental): Participants who had anti-programmed cell death-1 (PD-1)/programmed cell death ligand 1 (PD-L1) containing therapy but had progression of disease within ≤ 24 weeks from the start of treatment (primary resistance; PRI) will receive IV infusion of durvalumab 1500 mg Q4W in combination with oral olaparib 300 mg (2 × 150 mg) tablets BD until disease progression is confirmed.
  Interventions: Drug: Durvalumab; Drug: Olaparib
- Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg (Experimental): Participants who had progressive disease > 24 weeks from the start of anti PD-1/PD-L1 containing therapy while still on that treatment (acquired resistance; ACQ) will receive IV infusion of durvalumab 1500 mg Q4W in combination with oral olaparib 300 mg (2 × 150 mg) tablets BD until disease progression is confirmed.
  Interventions: Drug: Durvalumab; Drug: Olaparib
- Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg (Experimental): Participants who had anti-PD-1/PD-L1 containing therapy but had progression of disease within ≤ 24 weeks from the start of treatment (PRI) will receive IV infusion of AZD9150 (danvatirsen) 200 mg as loading dose on Days 1, 3, 5 of Cycle 0 (7-day-lead-in period). Thereafter, participants will receive AZD9150 200 mg every week (QW) on Days 1, 8, 15, and 22 of each 28-day cycle in combination with IV infusion of durvalumab 1500 mg Q4W, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
  Interventions: Drug: Durvalumab; Drug: Danvatirsen
- Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg (Experimental): Participants who had progressive disease > 24 weeks from the start of anti PD-1/PD-L1 containing therapy while still on that treatment (ACQ) will receive IV infusion of AZD9150 (danvatirsen) 200 mg as loading dose on Days 1, 3, 5 of Cycle 0 (7-day-lead-in period). Thereafter, participants will receive AZD9150 200 mg every week (QW) on Days 1, 8, 15, and 22 of each 28-day cycle in combination with IV infusion of durvalumab 1500 mg Q4W, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
  Interventions: Drug: Durvalumab; Drug: Danvatirsen
- Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg (Experimental): Participants who are ataxia telangiectasia mutated (ATM)-deficiecy will receive oral AZD6738 240 mg tablet BD for 7 days in Cycle 0 (Days 1 to 7). Thereafter, participants will receive IV infusion of durvalumab 1500 mg Q4W in combination with oral AZD6738 240 mg tablet BD in each cycle between Days 22 and 28 in each 28-day cycle, until objective radiological disease progression, however, participants may continue treatment if benefiting from treatment in the investigator opinion or did not meet any other discontinuation criteria.
  Interventions: Drug: Durvalumab; Drug: Ceralasertib
- Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg (Experimental): Participants who had anti-PD-1/PD-L1 containing therapy but had progression of disease within ≤ 24 weeks from the start of treatment (PRI) will receive oral AZD6738 240 mg tablet BD for 7 days in Cycle 0 (Days 1 to 7). Thereafter, participants will receive IV infusion of durvalumab 1500 mg Q4W in combination with oral AZD6738 240 mg tablet BD between Days 22 and 28 in each 28-day cycle, until objective radiological disease progression, however, participants may continue treatment if benefiting from treatment in the investigator opinion or did not meet any other discontinuation criteria.
  Interventions: Drug: Durvalumab; Drug: Ceralasertib
- Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg (Experimental): Participants who had progressive disease > 24 weeks from the start of anti PD-1/PD-L1 containing therapy while still on that treatment (ACQ) will receive oral AZD6738 240 mg tablet BD for 7 days in Cycle 0 (Days 1 to 7). Thereafter, participants will receive IV infusion of durvalumab 1500 mg Q4W in combination with oral AZD6738 240 mg tablet BD between Days 22 and 28 in each 28-day cycle, until objective radiological disease progression, however, participants may continue treatment if benefiting from treatment in the investigator opinion or did not meet any other discontinuation criteria.
  Interventions: Drug: Durvalumab; Drug: Ceralasertib
- Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg (Experimental): Participants with detectable genetic amplifications in rapamycin-insensitive companion of mechanistic target of rapamycin complex-2 (RICTOR) will receive IV infusion of durvalumab 1500 mg Q4W in combination with oral vistusertib 125 mg tablets BD on an intermittent dosing schedule of 2 days on, 5 days off, until objective radiological disease progression, however, participants may continue treatment if benefiting from treatment in the investigator opinion or did not meet any other discontinuation criteria.
  Interventions: Drug: Durvalumab; Drug: Vistusertib
- Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg (Experimental): Participants with high expression of cluster of differentiation 73 (CD73) will receive IV infusion of oleclumab 3000 mg every 2 weeks (Q2W) for 2 cycles and then Q4W thereafter in combination with IV infusion of durvalumab 1500 mg Q4W, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
  Interventions: Drug: Durvalumab; Drug: Oleclumab
- Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg (Experimental): Participants who had anti-PD-1/PD-L1 containing therapy but had progression of disease within ≤ 24 weeks from the start of treatment (PRI) will receive IV infusion of oleclumab 3000 mg Q2W for 2 cycles and then Q4W thereafter in combination with IV infusion of durvalumab 1500 mg Q4W, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
  Interventions: Drug: Durvalumab; Drug: Oleclumab
- Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg (Experimental): Participants who had progressive disease > 24 weeks from the start of anti PD-1/PD-L1 containing therapy while still on that treatment (ACQ) will receive IV infusion of oleclumab 3000 mg Q2W for 2 cycles and then Q4W thereafter in combination with IV infusion of durvalumab 1500 mg Q4W, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
  Interventions: Drug: Durvalumab; Drug: Oleclumab
- Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab deruxtecan 5.4mg/kg (Experimental): Participants whose tumours express human epidermal growth factor receptor 2 (HER2) mutations will receive IV infusion of trastuzumab deruxtecan (T-DXd) 5.4 mg/kg every 3 weeks (Q3W) in combination with IV infusion of durvalumab 1120 mg Q3W, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
  Interventions: Drug: Durvalumab; Drug: Trastuzumab deruxtecan
- Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab deruxtecan 5.4mg/kg (Experimental): Participants whose tumours harbour selected HER2 mutations will receive IV infusion of T-DXd 5.4 mg/kg Q3W in combination with IV infusion of durvalumab 1120 mg Q3W, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
  Interventions: Drug: Durvalumab; Drug: Trastuzumab deruxtecan
- Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg (Experimental): Participants who had progressive disease > 24 weeks from the start of anti PD-1/PD-L1 containing therapy while still on that treatment (ACQ) will receive IV infusion of durvalumab 1500 mg Q4W in combination with oral cediranib (AZD2171) 20 mg tablets daily for 5 days on, 2 days off (starting on Cycle 1 Day 1 of durvalumab), until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
  Interventions: Drug: Durvalumab; Drug: Cediranib
- Module 8 Cohort A.8.ATM: Ceralasertib 240 mg (Experimental): Participants who are ATM-deficient or with detectable aberrations in the ATM gene will receive oral ceralasertib (AZD6738) 240 mg tablets BD from Day 1 to Day 14 of each 28-day cycle, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
  Interventions: Drug: Ceralasertib
- Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg (Experimental): Participants who had anti-PD-1/PD-L1 containing therapy but had progression of disease within ≤ 24 weeks from the start of treatment (PRI) will receive IV infusion of durvalumab 1500 mg Q4W in combination with oral ceralasertib (AZD6738) 240 mg tablets BD for 14 days from Day 15 to Day 28 of each 28-day cycle, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
  Interventions: Drug: Durvalumab; Drug: Ceralasertib
- Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg (Experimental): Participants who had progressive disease > 24 weeks from the start of anti PD-1/PD-L1 containing therapy while still on that treatment (ACQ) will receive IV infusion of durvalumab 1500 mg Q4W plus oral ceralasertib (AZD6738) 240 mg tablets BD for 14 days from Day 15 to Day 28 of each 28-day cycle, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
  Interventions: Drug: Durvalumab; Drug: Ceralasertib
- Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg (Experimental): Participants, independent of their molecular aberration status, will receive oral ceralasertib (AZD6738) 160 mg tablet BD for 7 days in Cycle 0 (Days 1 to 7). Thereafter, participants will receive IV infusion of durvalumab 1500 mg Q4W in combination with oral ceralasertib 160 mg tablet BD between Days 22 and 28 in each 28-day cycle, until objective radiological disease progression, however, participants may continue treatment if benefiting from treatment in the investigator opinion or did not meet any other discontinuation criteria.
  Interventions: Drug: Durvalumab; Drug: Ceralasertib
- Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg (Experimental): Participants, independent of their molecular aberration status, will receive oral ceralasertib (AZD6738) 240 mg tablet BD for 7 days in Cycle 0 (Days 1 to 7). Thereafter, participants will receive IV infusion of durvalumab 1500 mg Q4W in combination with oral ceralasertib 240 mg tablet BD between Days 22 and 28 in each 28-day cycle, until objective radiological disease progression, however, participants may continue treatment if benefiting from treatment in the investigator opinion or did not meet any other discontinuation criteria.
  Interventions: Drug: Durvalumab; Drug: Ceralasertib
- Module 11 Cohort C.11.240: AZD6738 240 mg (Experimental): Participants, independent of their molecular aberration status, will receive oral AZD6738 tablet 240 mg for 7 days (Days 1 to 7) in each 28-day cycle until objective radiological disease progression, however, participants may continue treatment if benefiting from treatment in the investigator opinion or did not meet any other discontinuation criteria.
  Interventions: Drug: Ceralasertib

INTERVENTIONS:
Drug: Durvalumab — Participants will receive IV infusion of durvalumab as stated in arm description.
  Arms: Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg; Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg; Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg; Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg; Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg; Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg; Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg; Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg; Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg; Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg; Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg; Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg; Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg; Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg; Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg; Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab deruxtecan 5.4mg/kg; Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab deruxtecan 5.4mg/kg; Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg; Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg; Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg
Drug: Danvatirsen — Participants will receive IV infusion of danvatirsen as stated in arm description.
  Other Names: AZD9150
  Arms: Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg; Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg
Drug: Ceralasertib — Participants will receive oral tablet of ceralasertib as stated in arm description.
  Other Names: AZD6738
  Arms: Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg; Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg; Module 11 Cohort C.11.240: AZD6738 240 mg; Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg; Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg; Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg; Module 8 Cohort A.8.ATM: Ceralasertib 240 mg; Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg; Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg
Drug: Vistusertib — Participants will receive oral tablets of vistusertib as stated in arm description.
  Arms: Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg
Drug: Olaparib — Participants will receive oral tablets of olaparib as stated in arm description.
  Arms: Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg; Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg; Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg; Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg
Drug: Oleclumab — Participants will receive IV infusion of oleclumab as stated in arm description.
  Arms: Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg; Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg; Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg
Drug: Trastuzumab deruxtecan — Participants will receive IV infusion of trastuzumab deruxtecan as stated in arm description.
  Other Names: T-DXd
  Arms: Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab deruxtecan 5.4mg/kg; Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab deruxtecan 5.4mg/kg
Drug: Cediranib — Participants will receive oral tablets of cediranib as stated in arm description.
  Other Names: AZD2171
  Arms: Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg

SUMMARY:
This is an open-label, multi-centre, umbrella Phase II study in participants with metastatic NSCLC who have progressed on an anti-PD-1/PD-L1 containing therapy. This study is modular in design, allowing initial assessment of the efficacy, safety, and tolerability of multiple treatment arms.

DETAILED DESCRIPTION:
This is an open-label, multi-centre, umbrella Phase II study in participants with metastatic non-small cell lung cancer (NSCLC) who have progressed on an anti-programmed cell death-1/anti-programmed cell death ligand 1 (anti-PD-1/PD-L1) containing therapy. This study is modular in design, consisting of a number of treatment cohorts, allowing evaluation of the efficacy, safety, and tolerability of multiple treatment arms. There is currently no established therapy for participants who have received immune checkpoint inhibitors and platinum-doublet therapies, and novel treatments are urgently needed.

This protocol has a modular design, with the potential for future treatment arms to be added via protocol amendment.

ELIGIBILITY:
Inclusion criteria:

* At least 18 years of age at the time of signing the informed consent form.
* Participant must have histologically or cytologically confirmed metastatic or locally advanced and recurrent non-small-cell lung cancer (NSCLC) which is progressing.
* Participants eligible for second- or later-line therapy, who must have received an anti-programmed cell death protein-1 (PD-1)/programmed death-ligand 1 (PD-L1) containing therapy and a platinum-doublet regimen for locally advanced or metastatic NSCLC either separately or in combination. Prior durvalumab is acceptable. The participant must have had disease progression on a prior line of anti-PD-1/PD-L1 therapy.
* Eastern Cooperative Oncology Group/World Health Organization (ECOG/WHO) performance status of 0 to 1, and a minimum life expectancy of 12 weeks.
* Participant must have at least 1 lesion that can be accurately measured. A previously irradiated lesion can be considered a target lesion if the lesion has clearly progressed.
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal participants.

Exclusion Criteria:

* Participants whose tumour samples have targetable alterations in epidermal growth factor receptor (EGFR) and/or anaplastic lymphoma kinase (ALK) at initial diagnosis are excluded. In addition, participants whose tumour samples are known to have targetable alterations in ROS1, BRAF, MET or RET, are to be excluded.
* Active or prior documented autoimmune or inflammatory disorders.
* Active infection including tuberculosis, hepatitis B (known positive hepatitis B virus [HBV] surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus (positive human immunodeficiency virus [HIV] 1/2 antibodies).
* Female participant who are pregnant or breastfeeding, or male or female participants of reproductive potential who are not willing to employ effective birth control.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients, or history of severe hypersensitivity reactions to other monoclonal antibodies.
* Participant has spinal cord compression or symptomatic brain metastases.
* Any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment. Participants may receive treatment with bisphosphonates or receptor activator of nuclear factor kappa-Β ligand (RANKL) inhibitors for the treatment of bone metastases.
* History of active primary immunodeficiency.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2026-09-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John Heymach, M.D, Ph.D, Principal Investigator — M.D. Anderson Cancer Center
Locations (39):
- United States (15):
  - Research Site, Duarte, California
  - Research Site, Fullerton, California
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Fairfax, Virginia
- Austria (3):
  - Research Site, Innsbruck
  - Research Site, Salzburg
  - Research Site, Vienna
- Canada (5):
  - Research Site, Edmonton, Alberta
  - Research Site, Brampton, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- France (4):
  - Research Site, Bordeaux
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Villejuif
- Germany (4):
  - Research Site, Berlin
  - Research Site, Esslingen a.N.
  - Research Site, Großhansdorf
  - Research Site, Heidelberg
- Israel (4):
  - Research Site, Haifa
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
- Research Site, Seoul, South Korea
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Besse B, Pons-Tostivint E, Park K, Hartl S, Forde PM, Hochmair MJ, Awad MM, Thomas M, Goss G, Wheatley-Price P, Shepherd FA, Florescu M, Cheema P, Chu QSC, Kim SW, Morgensztern D, Johnson ML, Cousin S, Kim DW, Moskovitz MT, Vicente D, Aronson B, Hobson R, Ambrose HJ, Khosla S, Reddy A, Russell DL, Keddar MR, Conway JP, Barrett JC, Dean E, Kumar R, Dressman M, Jewsbury PJ, Iyer S, Barry ST, Cosaert J, Heymach JV. Biomarker-directed targeted therapy plus durvalumab in advanced non-small-cell lung cancer: a phase 2 umbrella trial. Nat Med. 2024 Mar;30(3):716-729. doi: 10.1038/s41591-024-02808-y. Epub 2024 Feb 13. PMID 38351187
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6185C00001&attachmentIdentifier=73155d56-c95a-483f-9c56-630afd5df1e8&fileName=D6185c00001-SAP-v9.0_15Feb24.pdf&versionIdentifier=
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6185C00001&attachmentIdentifier=7d0cabb4-4573-443e-ab4f-1f9f777874f2&fileName=d6185c00001-csp-v14_Redacted.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6185C00001&attachmentIdentifier=35106804-b43c-4872-b55a-63b9b4465ba2&fileName=CSR_Synopsis_(Modules_1-11)_Redacted_PDF-A.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 45 centers in 8 countries (Austria, Canada, France, Germany, Israel, South Korea, Spain, and the United States).
Pre-assignment Details: A total of 529 participants were enrolled in this study.
Groups:
- Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg: Participants with detectable aberrations, mutation detected in a homologous recombination repair gene (HRRm) received IV infusion of durvalumab 1500 mg every 4 weeks (Q4W) in combination with oral olaparib 300 mg (2 × 150 mg) tablets twice a day (BD) until disease progression is confirmed.
- Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg: Participants with detectable aberrations in liver kinase B1 (LKB1) received IV infusion of durvalumab 1500 mg Q4W in combination with oral olaparib 300 mg (2 × 150 mg) tablets BD until disease progression is confirmed.
- Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg: Participants who had anti-programmed cell death-1 (PD-1)/programmed cell death ligand 1 (PD-L1) containing therapy but had progression of disease within ≤ 24 weeks from the start of treatment (primary resistance; PRI) received IV infusion of durvalumab 1500 mg Q4W in combination with oral olaparib 300 mg (2 × 150 mg) tablets BD until disease progression is confirmed.
- Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg: Participants who had progressive disease > 24 weeks from the start of anti PD-1/PD-L1 containing therapy while still on that treatment (acquired resistance; ACQ) received IV infusion of durvalumab 1500 mg Q4W in combination with oral olaparib 300 mg (2 × 150 mg) tablets BD until disease progression is confirmed.
- Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg: Participants who had anti-PD-1/PD-L1 containing therapy but had progression of disease within ≤ 24 weeks from the start of treatment (PRI) received IV infusion of AZD9150 (danvatirsen) 200 mg as loading dose on Days 1, 3, 5 of Cycle 0 (7-day-lead-in period). Thereafter, participants received AZD9150 200 mg every week (QW) on Days 1, 8, 15, and 22 of each 28-day cycle in combination with IV infusion of durvalumab 1500 mg Q4W, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
- Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg: Participants who had progressive disease > 24 weeks from the start of anti PD-1/PD-L1 containing therapy while still on that treatment (ACQ) received IV infusion of AZD9150 (danvatirsen) 200 mg as loading dose on Days 1, 3, 5 of Cycle 0 (7-day-lead-in period). Thereafter, participants received AZD9150 200 mg every week (QW) on Days 1, 8, 15, and 22 of each 28-day cycle in combination with IV infusion of durvalumab 1500 mg Q4W, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
- Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg: Participants who are ataxia telangiectasia mutated (ATM)-deficiecy received oral AZD6738 240 mg tablet BD for 7 days in Cycle 0 (Days 1 to 7). Thereafter, participants received IV infusion of durvalumab 1500 mg Q4W in combination with oral AZD6738 240 mg tablet BD in each cycle between Days 22 and 28 in each 28-day cycle, until objective radiological disease progression, however, participants may continue treatment if benefiting from treatment in the investigator opinion or did not meet any other discontinuation criteria.
- Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg: Participants who had anti-PD-1/PD-L1 containing therapy but had progression of disease within ≤ 24 weeks from the start of treatment (PRI) received oral AZD6738 240 mg tablet BD for 7 days in Cycle 0 (Days 1 to 7). Thereafter, participants received IV infusion of durvalumab 1500 mg Q4W in combination with oral AZD6738 240 mg tablet BD between Days 22 and 28 in each 28-day cycle, until objective radiological disease progression, however, participants may continue treatment if benefiting from treatment in the investigator opinion or did not meet any other discontinuation criteria.
- Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg: Participants who had progressive disease > 24 weeks from the start of anti PD-1/PD-L1 containing therapy while still on that treatment (ACQ) received oral AZD6738 240 mg tablet BD for 7 days in Cycle 0 (Days 1 to 7). Thereafter, participants received IV infusion of durvalumab 1500 mg Q4W in combination with oral AZD6738 240 mg tablet BD between Days 22 and 28 in each 28-day cycle, until objective radiological disease progression, however, participants may continue treatment if benefiting from treatment in the investigator opinion or did not meet any other discontinuation criteria.
- Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg: Participants with detectable genetic amplifications in rapamycin-insensitive companion of mechanistic target of rapamycin complex-2 (RICTOR) received IV infusion of durvalumab 1500 mg Q4W in combination with oral vistusertib 125 mg tablets BD on an intermittent dosing schedule of 2 days on, 5 days off, until objective radiological disease progression, however, participants may continue treatment if benefiting from treatment in the investigator opinion or did not meet any other discontinuation criteria.
- Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg: Participants with high expression of cluster of differentiation 73 (CD73) received IV infusion of oleclumab 3000 mg every 2 weeks (Q2W) for 2 cycles and then Q4W thereafter in combination with IV infusion of durvalumab 1500 mg Q4W, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
- Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg: Participants who had anti-PD-1/PD-L1 containing therapy but had progression of disease within ≤ 24 weeks from the start of treatment (PRI) received IV infusion of oleclumab 3000 mg Q2W for 2 cycles and then Q4W thereafter in combination with IV infusion of durvalumab 1500 mg Q4W, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
- Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg: Participants who had progressive disease > 24 weeks from the start of anti PD-1/PD-L1 containing therapy while still on that treatment (ACQ) received IV infusion of oleclumab 3000 mg Q2W for 2 cycles and then Q4W thereafter in combination with IV infusion of durvalumab 1500 mg Q4W, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
- Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg: Participants whose tumours express human epidermal growth factor receptor 2 (HER2) mutations received IV infusion of trastuzumab deruxtecan (T-DXd) 5.4 mg/kg every 3 weeks (Q3W) in combination with IV infusion of durvalumab 1120 mg Q3W, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
- Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg: Participants whose tumours harbour selected HER2 mutations received IV infusion of T-DXd 5.4 mg/kg Q3W in combination with IV infusion of durvalumab 1120 mg Q3W, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
- Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg: Participants who had progressive disease > 24 weeks from the start of anti PD-1/PD-L1 containing therapy while still on that treatment (ACQ) received IV infusion of durvalumab 1500 mg Q4W in combination with oral cediranib (AZD2171) 20 mg tablets daily for 5 days on, 2 days off (starting on Cycle 1 Day 1 of durvalumab), until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
- Module 8 Cohort A.8.ATM: Ceralasertib 240 mg: Participants who are ATM-deficient or with detectable aberrations in the ATM gene received oral ceralasertib (AZD6738) 240 mg tablets BD from Day 1 to Day 14 of each 28-day cycle, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
- Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg: Participants who had anti-PD-1/PD-L1 containing therapy but had progression of disease within ≤ 24 weeks from the start of treatment (PRI) received IV infusion of durvalumab 1500 mg Q4W in combination with oral ceralasertib (AZD6738) 240 mg tablets BD for 14 days from Day 15 to Day 28 of each 28-day cycle, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
- Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg: Participants who had progressive disease > 24 weeks from the start of anti PD-1/PD-L1 containing therapy while still on that treatment (ACQ) received IV infusion of durvalumab 1500 mg Q4W plus oral ceralasertib (AZD6738) 240 mg tablets BD for 14 days from Day 15 to Day 28 of each 28-day cycle, until objective radiological disease progression, as long as, in the investigator's opinion, they were benefiting from treatment and did not meet any other discontinuation criteria.
- Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg: Participants, independent of their molecular aberration status, received oral ceralasertib (AZD6738) 160 mg tablet BD for 7 days in Cycle 0 (Days 1 to 7). Thereafter, participants received IV infusion of durvalumab 1500 mg Q4W in combination with oral ceralasertib 160 mg tablet BD between Days 22 and 28 in each 28-day cycle, until objective radiological disease progression, however, participants may continue treatment if benefiting from treatment in the investigator opinion or did not meet any other discontinuation criteria.
- Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg: Participants, independent of their molecular aberration status, received oral ceralasertib (AZD6738) 240 mg tablet BD for 7 days in Cycle 0 (Days 1 to 7). Thereafter, participants received IV infusion of durvalumab 1500 mg Q4W in combination with oral ceralasertib 240 mg tablet BD between Days 22 and 28 in each 28-day cycle, until objective radiological disease progression, however, participants may continue treatment if benefiting from treatment in the investigator opinion or did not meet any other discontinuation criteria.
- Module 11 Cohort C.11.240: AZD6738 240 mg: Participants, independent of their molecular aberration status, received oral AZD6738 tablet 240 mg for 7 days (Days 1 to 7) in each 28-day cycle until objective radiological disease progression, however, participants may continue treatment if benefiting from treatment in the investigator opinion or did not meet any other discontinuation criteria.
Period: Overall Study
Arm/Group | Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg | Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg | Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg | Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg | Module 8 Cohort A.8.ATM: Ceralasertib 240 mg | Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg | Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 11 Cohort C.11.240: AZD6738 240 mg
Started | 21 | 21 | 22 | 23 | 23 | 22 | 31 | 38 | 58 | 1 | 23 | 9 | 25 | 23 | 20 | 22 | 15 | 19 | 24 | 34 | 17 | 38
Completed | 2 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Not Completed | 19 | 21 | 20 | 23 | 22 | 20 | 31 | 38 | 57 | 0 | 23 | 8 | 25 | 23 | 20 | 22 | 15 | 19 | 24 | 33 | 17 | 36
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 18 | 18 | 20 | 21 | 20 | 16 | 28 | 35 | 47 | 0 | 19 | 6 | 20 | 22 | 17 | 18 | 12 | 15 | 16 | 27 | 14 | 27
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 1
Not completed — Other | 1 | 2 | 0 | 1 | 1 | 0 | 2 | 1 | 8 | 0 | 3 | 1 | 3 | 1 | 1 | 3 | 3 | 3 | 7 | 4 | 1 | 4
Not completed — Continuing study off treatment at data cut-off | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Intention to treat (ITT) analysis population included all enrolled participants who received at least 1 dose of the study drug and were analyzed according to their assigned cohort and planned treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg | Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg | Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg | Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg | Module 8 Cohort A.8.ATM: Ceralasertib 240 mg | Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg | Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 11 Cohort C.11.240: AZD6738 240 mg | Total
Number analyzed (Participants) | 21 | 21 | 22 | 23 | 23 | 22 | 31 | 38 | 58 | 1 | 23 | 9 | 25 | 23 | 20 | 22 | 15 | 19 | 24 | 34 | 17 | 38 | 529
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (10.4) | 60.2 (11.6) | 60.9 (7.6) | 66.5 (8.6) | 63.7 (9.8) | 64.1 (9.5) | 61.2 (8.2) | 62.2 (8.8) | 62.7 (9.4) | NA (NA) — Mean was not reported due to concern with participant's confidentiality. Standard deviation is not calculated as only one participant is involved in Module 4. | 60.4 (10.2) | 61.9 (7.6) | 66.2 (8.6) | 62.7 (11.1) | 61.5 (12.8) | 65.8 (8.8) | 66.7 (8.2) | 61.1 (8.5) | 67.4 (11.5) | 62.4 (8.4) | 64.1 (10.9) | 62.6 (8.4) | 63.0 (9.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 8 | 9 | 12 | 8 | 11 | 11 | 15 | 10 | 17 | 0 | 11 | 7 | 9 | 8 | 11 | 5 | 5 | 5 | 10 | 9 | 4 | 13 | 198
  Male | 13 | 12 | 10 | 15 | 12 | 11 | 16 | 28 | 41 | 0 | 12 | 2 | 16 | 15 | 9 | 17 | 10 | 14 | 14 | 25 | 13 | 25 | 330
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Not Hispanic or Latino | 21 | 20 | 22 | 23 | 21 | 22 | 29 | 36 | 55 | 0 | 22 | 9 | 23 | 21 | 19 | 21 | 15 | 19 | 24 | 34 | 17 | 38 | 511
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 2 | 3 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 0 | 8 | 11 | 1 | 6 | 0 | 8 | 6 | 0 | 1 | 0 | 7 | 5 | 4 | 3 | 1 | 4 | 4 | 6 | 3 | 5 | 87
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 12
  White | 15 | 19 | 13 | 11 | 15 | 14 | 23 | 15 | 33 | 0 | 15 | 9 | 13 | 15 | 13 | 16 | 12 | 9 | 15 | 21 | 11 | 33 | 340
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 1 | 1 | 5 | 0 | 8 | 13 | 16 | 1 | 6 | 0 | 5 | 3 | 1 | 2 | 2 | 6 | 5 | 7 | 3 | 0 | 89

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response Per Response Evaluation Criteria in Solid Tumours Version 1.1 (RECIST v1.1)
Description: Objective response was defined as participants with a confirmed investigator-assessed response complete response (CR) or partial response (PR) based on RECIST v 1.1. The CR is defined as disappearance of all target (TL) and non-target lesions (NTL), and any pathological lymph node (whether target or nontarget) must have reduction in short axis to <10 mm. The PR is defined as at least a 30% decrease in the sum of the diameters of TLs, taking as reference the baseline sum diameters, as long as criteria for progressive disease (PD) are not met. Confirmation of CR and PR is required by a repeat, consecutive assessment no less than 4 weeks from date of first documentation. Percentage of participants with objective response was reported.
Time Frame: Baseline (<=28 days before treatment), then every 6 weeks for 24 weeks from Cycle 1 Day 1, then every 8 weeks (every 9 weeks in Module 6) until disease progression or 90 days after study drug discontinuation (approximately 2 years)
Population: Evaluable for response population included all dosed participants who had measurable disease at baseline and who were analyzed according to their assigned cohort and planned treatment.
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg | Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg | Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg | Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg | Module 8 Cohort A.8.ATM: Ceralasertib 240 mg | Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg | Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 11 Cohort C.11.240: AZD6738 240 mg
Number analyzed (Participants) | 21 | 21 | 22 | 23 | 23 | 22 | 31 | 37 | 58 | 1 | 23 | 9 | 25 | 23 | 20 | 22 | 15 | 18 | 24 | 34 | 17 | 38
Percentage of Participants | 9.5 [2.6 to 23.4] | 4.8 [0.5 to 17.3] | 0 [0.0 to 9.9] | 4.3 [0.5 to 15.9] | 0 [0.0 to 9.5] | 0 [0.0 to 9.9] | 25.8 [15.7 to 38.5] | 8.1 [3.0 to 17.2] | 8.6 [4.3 to 15.4] | NA [NA to NA] — No efficacy data were collected as the module was prematurely discontinued by the sponsor for strategic reasons. At the time of decision to discontinue the module, only a single participant had received treatment, and only safety data were collected on that participant. | 4.3 [0.5 to 15.9] | 0 [0.0 to 22.6] | 4.0 [0.4 to 14.7] | 21.7 [11.0 to 36.6] | 35.0 [20.7 to 51.8] | 22.7 [11.5 to 38.1] | 0 [0.0 to 14.2] | 16.7 [6.3 to 33.4] | 8.3 [2.2 to 20.7] | 0 [0.0 to 6.5] | 11.8 [3.2 to 28.4] | 2.6 [0.3 to 9.9]

2. Secondary Outcome: Overall Survival (OS)
Description: The OS is defined as the time from the first dose of any study drug until death due to any cause regardless of whether the participant withdraws from study treatment or receives subsequent cancer therapy. The overall survival was analyzed using the Kaplan-Meier method.
Time Frame: Every 3 months after safety follow-up visit (90 days after study drug discontinuation) until planned database lock for a module (either 12 months after last participant has started treatment or when 75% of participants died) (approximately up to 2 years)
Population: as for baseline characteristics
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg | Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg | Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg | Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg | Module 8 Cohort A.8.ATM: Ceralasertib 240 mg | Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg | Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 11 Cohort C.11.240: AZD6738 240 mg
Number analyzed (Participants) | 21 | 21 | 22 | 23 | 23 | 22 | 31 | 38 | 58 | 1 | 23 | 9 | 25 | 23 | 20 | 22 | 15 | 19 | 24 | 34 | 17 | 38
Months | 9.63 [5.26 to 15.97] | 5.75 [5.29 to 10.84] | 7.16 [4.93 to 10.28] | 15.51 [9.33 to 20.86] | 6.01 [3.55 to 6.51] | 11.20 [9.72 to 12.55] | 15.80 [14.16 to 22.80] | 10.22 [5.82 to 11.30] | 11.37 [9.13 to 15.80] | NA [NA to NA] — No efficacy data were collected as the module was prematurely discontinued by the sponsor for strategic reasons. At the time of decision to discontinue the module, only a single participant had received treatment, and only safety data were collected on that participant. | 10.97 [7.59 to 15.74] | 7.06 [4.90 to 11.99] | 12.78 [7.39 to 20.96] | 9.53 [6.57 to 12.42] | 10.61 [8.90 to 20.60] | 14.19 [11.86 to 19.88] | 14.23 [6.08 to 17.18] | 7.95 [5.59 to 8.64] | 12.91 [7.39 to 20.50] | 5.95 [4.01 to 10.05] | 7.03 [4.37 to 12.71] | 6.60 [5.85 to 9.13]

3. Secondary Outcome: Progression-Free Survival (PFS) Per RECIST v1.1
Description: The PFS is defined as time from first dose of any study drug until date of objective disease progression (PD) per RECIST v1.1 or death by any cause, regardless of whether the participant withdraws from study therapy or receives another anti-cancer therapy prior to progression. The PD is defined as a >= 20% increase in the sum of diameters of TLs and an absolute increase of >= 5mm, taking as reference the smallest sum of diameters since treatment started including the baseline sum of diameters, or unequivocal progression of existing NTL. The PFS was analyzed using the Kaplan-Meier method
Time Frame: as for outcome 2
Population: The ITT analysis population included all enrolled participants who received at least 1 dose of the study drug and were analyzed according to their assigned cohort and planned treatment.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg | Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg | Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg | Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg | Module 8 Cohort A.8.ATM: Ceralasertib 240 mg | Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg | Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 11 Cohort C.11.240: AZD6738 240 mg
Number analyzed (Participants) | 21 | 21 | 22 | 23 | 23 | 22 | 31 | 38 | 58 | 1 | 23 | 9 | 25 | 23 | 20 | 22 | 15 | 19 | 24 | 34 | 17 | 38
Months | 2.79 [1.41 to 5.26] | 1.41 [1.38 to 1.81] | 3.38 [2.10 to 4.93] | 4.17 [2.69 to 4.37] | 1.68 [1.64 to 2.99] | 3.09 [2.83 to 6.14] | 7.43 [5.59 to 9.43] | 2.96 [1.91 to 3.09] | 4.21 [3.02 to 4.96] | NA [NA to NA] — No efficacy data were collected as the module was prematurely discontinued by the sponsor for strategic reasons. At the time of decision to discontinue the module, only a single participant had received treatment, and only safety data were collected on that participant. | 1.61 [1.41 to 2.76] | 1.41 [1.35 to 1.81] | 2.69 [1.74 to 4.17] | 2.83 [2.33 to 5.45] | 5.52 [5.32 to 5.72] | 4.17 [2.56 to 9.36] | 3.42 [2.14 to 7.62] | 1.48 [1.41 to 2.23] | 3.68 [2.83 to 7.33] | 1.68 [1.61 to 2.56] | 2.00 [1.71 to 2.79] | 2.86 [2.73 to 3.02]

4. Secondary Outcome: Best Percentage Change From Baseline in Tumour Size
Description: The best percentage change in tumour size from baseline i.e. the maximum reduction from baseline or the minimum increase from baseline in absence of a reduction from baseline based on all post baseline assessments is reported. Tumour size is sum of the longest diameters (or short axis measurements for lymph nodes) of the target lesions. Baseline was defined as last evaluable assessment prior to starting treatment. The percentage change in target lesion tumour size at each week X for which data are available was obtained for each participant taking the difference between the sum of the target lesions at each week X and the sum of the target lesions at baseline divided by the sum of the target lesions at baseline multiplied by 100 (i.e. [week X - baseline]/baseline * 100).
Time Frame: Baseline (<=28 days prior to starting treatment) then every 6 weeks for first 24 weeks relative to the date of first dose/combination therapy (Cycle 1 Day 1), then every 8 weeks (except Module 6)/9 weeks (Module 6) thereafter (approximately up to 2 years)
Population: Evaluable for response population included all dosed participants who had measurable disease at baseline and who were analyzed according to their assigned cohort and planned treatment. Number of participants analyzed (N) denotes the number of participants evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent Change in Tumor Size
Arm/Group | Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg | Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg | Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg | Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg | Module 8 Cohort A.8.ATM: Ceralasertib 240 mg | Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg | Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 11 Cohort C.11.240: AZD6738 240 mg
Number analyzed (Participants) | 21 | 21 | 22 | 23 | 23 | 21 | 31 | 37 | 58 | 1 | 23 | 9 | 25 | 23 | 20 | 22 | 15 | 17 | 23 | 34 | 17 | 38
Percent Change in Tumor Size | -0.79 (25.706) | 10.24 (25.197) | 7.19 (21.082) | -3.55 (20.879) | 16.36 (20.732) | 3.06 (19.015) | -10.12 (33.560) | 3.39 (29.846) | -0.03 (29.952) | NA (NA) — No efficacy data were collected as the module was prematurely discontinued by the sponsor for strategic reasons. At the time of decision to discontinue the module, only a single participant had received treatment, and only safety data were collected on that participant. | 15.15 (24.412) | 19.55 (21.537) | 6.62 (29.231) | -14.15 (35.815) | -32.22 (35.655) | -8.62 (38.546) | -6.40 (17.207) | 8.96 (46.410) | -2.59 (27.957) | 15.88 (34.908) | 19.74 (43.830) | -1.14 (22.354)

5. Secondary Outcome: Percentage of Participants With Disease Control (DC) Per RECIST v1.1
Description: Module (M) 1, 4, 5, 6, 7, 8, 9, 11: DCR at 12 and 24 weeks is defined as percentage of participants who have best overall response (BoR) of CR or PR in first 13/25 weeks, respectively, post start of any study drug or with duration of SD for at least 11/23 weeks, respectively, after start of any study drug. M2, M3, M10: DCR at 12 and 24 weeks is defined as percentage of participants who have BoR of CR or PR within first 100 days (M2, M3, M10) or 184 days (M2, M3, M10) after start of any study drug, or have SD lasting at least 86 days (M2)/82 days (M3, M10), respectively, or 170 days (M2)/166 days (M3, M10), respectively, post start of any study drug. CR is defined as disappearance of all TL and NTLs, and any pathological lymph node (whether target or nontarget) must have reduction in short axis to <10 mm. PR is defined as at least 30% decrease in sum of diameters of TLs, taking as reference baseline sum diameters, as long as criteria for PD are not met.
Time Frame: At 12 and 24 weeks after the start of study drug
Population: as for outcome 1
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg | Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg | Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg | Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg | Module 8 Cohort A.8.ATM: Ceralasertib 240 mg | Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg | Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 11 Cohort C.11.240: AZD6738 240 mg
Number analyzed (Participants) | 21 | 21 | 22 | 23 | 23 | 22 | 31 | 37 | 58 | 1 | 23 | 9 | 25 | 23 | 20 | 22 | 15 | 18 | 24 | 34 | 17 | 38
Percentage of Participants
  At 12 weeks | 38.1 [23.6 to 54.4] | 9.5 [2.6 to 23.4] | 45.5 [30.5 to 61.1] | 52.2 [37.0 to 67.0] | 13.0 [4.9 to 26.8] | 40.9 [26.4 to 56.8] | 67.7 [54.7 to 78.9] | 54.1 [42.3 to 65.5] | 58.6 [49.4 to 67.4] | NA [NA to NA] — No efficacy data were collected as the module was prematurely discontinued by the sponsor for strategic reasons. At the time of decision to discontinue the module, only a single participant had received treatment, and only safety data were collected on that participant. | 34.8 [21.4 to 50.3] | 22.2 [6.1 to 49.0] | 56.0 [41.3 to 69.9] | 56.5 [41.1 to 71.0] | 70.0 [53.3 to 83.4] | 63.6 [47.7 to 77.5] | 60.0 [40.4 to 77.4] | 22.2 [10.1 to 39.6] | 58.3 [43.3 to 72.3] | 32.4 [21.7 to 44.7] | 41.2 [24.6 to 59.4] | 60.5 [48.8 to 71.3]
  At 24 weeks | 19.0 [8.6 to 34.5] | 9.5 [2.6 to 23.4] | 13.6 [5.1 to 27.9] | 26.1 [14.3 to 41.3] | 0 [0.0 to 9.5] | 27.3 [15.0 to 43.0] | 58.1 [45.0 to 70.3] | 27.0 [17.5 to 38.5] | 34.5 [26.2 to 43.7] | NA [NA to NA] — No efficacy data were collected as the module was prematurely discontinued by the sponsor for strategic reasons. At the time of decision to discontinue the module, only a single participant had received treatment, and only safety data were collected on that participant. | 8.7 [2.3 to 21.5] | 11.1 [1.2 to 36.8] | 24.0 [13.1 to 38.3] | 34.8 [21.4 to 50.3] | 60.0 [43.3 to 75.1] | 45.5 [30.5 to 61.1] | 40.0 [22.6 to 59.6] | 16.7 [6.3 to 33.4] | 33.3 [20.5 to 48.4] | 17.6 [9.5 to 28.9] | 23.5 [10.7 to 41.6] | 26.3 [17.0 to 37.6]

6. Secondary Outcome: Duration of Response (DoR) Per RECIST v1.1
Description: The DoR is defined as the time from the first documented confirmed response (CR or PR) until the first documented PD or death in the absence of disease progression. The CR is defined as disappearance of all TLs and NTLs, and any pathological lymph node (whether target or nontarget) must have reduction in short axis to <10 mm. The PR is defined as at least a 30 decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters, as long as criteria for PD are not met. The PD is defined as a >=20% increase in the sum of diameters of TLs and an absolute increase of >=5mm, taking as reference the smallest sum of diameters since treatment started including the baseline sum of diameters, or unequivocal progression of existing NTL. The DoR was analyzed using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: Evaluable for response population included all dosed participants who had measurable disease at baseline and who were analyzed according to their assigned cohort and planned treatment. The DoR was assessed for only those participants who had OR. Here, number of participants denotes those participants who had OR (confirmed CR or PR).
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg | Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg | Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg | Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg | Module 8 Cohort A.8.ATM: Ceralasertib 240 mg | Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg | Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 11 Cohort C.11.240: AZD6738 240 mg
Number analyzed (Participants) | 2 | 1 | 0 | 1 | 0 | 0 | 8 | 3 | 5 | 0 | 1 | 0 | 1 | 5 | 7 | 5 | 0 | 3 | 2 | 0 | 2 | 1
Months | NA [NA to NA] — Number of responders were less than 3, hence median and the quartiles of were not calculated. | NA [NA to NA] — Number of responders were less than 3, hence median and the quartiles were not calculated. |  | NA [NA to NA] — Number of responders were less than 3, hence median and the quartiles were not calculated. |  |  | 6.57 [5.95 to 13.24] | 10.45 [3.94 to 10.45] | 34.83 [7.85 to 34.83] |  | NA [NA to NA] — Number of responders were less than 3, hence median and the quartiles were not calculated. |  | NA [NA to NA] — Number of responders were less than 3, hence median and the quartiles were not calculated. | 6.60 [4.17 to NA] — Third quartile was not calculated as percentage of events associated with that quartile was not met by end of study follow-up. | 4.14 [2.79 to 5.32] | 11.10 [6.18 to 19.68] |  | NA [1.87 to NA] — Median and third quartile were not calculated as percentage of events associated with that median and quartile were not met by end of study follow-up. | NA [NA to NA] — Number of responders were less than 3, hence median and the quartiles were not calculated. |  | NA [NA to NA] — Number of responders were less than 3, hence median and the quartiles were not calculated. | NA [NA to NA] — Number of responders were less than 3, hence median and the quartiles were not calculated.

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 thorugh 58.6 months (maximum observed duration)
Population: Safety analysis set included participants who received at least 1 dose of study drug and who were analyzed according to the actual treatment received and corresponding assigned cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg | Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg | Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg | Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg | Module 8 Cohort A.8.ATM: Ceralasertib 240 mg | Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg | Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 11 Cohort C.11.240: AZD6738 240 mg
Number analyzed (Participants) | 21 | 21 | 22 | 23 | 23 | 22 | 31 | 38 | 58 | 1 | 23 | 9 | 25 | 23 | 20 | 22 | 15 | 19 | 24 | 34 | 17 | 38
Participants
  Any TEAEs | 20 | 19 | 20 | 21 | 23 | 20 | 31 | 35 | 56 | 1 | 21 | 5 | 22 | 23 | 20 | 21 | 15 | 17 | 24 | 32 | 16 | 38
  Any TESAEs | 10 | 7 | 8 | 7 | 12 | 8 | 11 | 11 | 17 | 0 | 7 | 1 | 6 | 10 | 10 | 7 | 7 | 7 | 13 | 12 | 1 | 17

8. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs
Description: Number of participants with abnormal clinical laboratory parameters reported as TEAEs are reported. Abnormal clinical laboratory parameters defined as any abnormal finding during analysis of hematology, clinical chemistry, and urinalysis.
Time Frame: Day 1 thorugh 58.6 months (maximum observed duration)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg | Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg | Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg | Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg | Module 8 Cohort A.8.ATM: Ceralasertib 240 mg | Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg | Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 11 Cohort C.11.240: AZD6738 240 mg
Number analyzed (Participants) | 21 | 21 | 22 | 23 | 23 | 22 | 31 | 38 | 58 | 1 | 23 | 9 | 25 | 23 | 20 | 22 | 15 | 19 | 24 | 34 | 17 | 38
Participants
  Anaemia | 7 | 7 | 5 | 7 | 4 | 4 | 10 | 9 | 19 | 0 | 1 | 1 | 3 | 7 | 12 | 1 | 12 | 8 | 12 | 5 | 7 | 15
  Thrombocytopenia | 1 | 1 | 0 | 0 | 4 | 6 | 4 | 2 | 4 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 5 | 10 | 1 | 2 | 2
  Hyponatraemia | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 7 | 0 | 0 | 0 | 1 | 2 | 5 | 2 | 2 | 2 | 2 | 3 | 1 | 4
  Hypokalaemia | 4 | 2 | 1 | 1 | 2 | 1 | 2 | 0 | 5 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 3 | 2 | 4 | 0 | 0 | 2
  Aspartate aminotransferase increased | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 1 | 3 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 0 | 4 | 0 | 2 | 2
  Blood creatinine increased | 2 | 1 | 3 | 1 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 2 | 1 | 2 | 0 | 0 | 2
  Hypoalbuminaemia | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 5 | 0 | 2 | 0 | 0 | 0 | 1 | 5
  Platelet count decreased | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 4 | 1 | 6 | 0 | 0 | 1
  Alanine aminotransferase increased | 0 | 0 | 0 | 0 | 3 | 5 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 3
  C-reactive protein increased | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 4
  Hypomagnesaemia | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 3
  Hyperglycaemia | 2 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 1
  Lymphocyte count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 3 | 2 | 2 | 0 | 1 | 0 | 0 | 1
  Lipase increased | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 1 | 2 | 0 | 0 | 1
  Neutrophil count decreased | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 2 | 1 | 2 | 0 | 0 | 1
  Blood alkaline phosphatase increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 2 | 0 | 0 | 1
  Hypophosphataemia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 4
  Neutropenia | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 2
  White blood cell count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 4 | 1 | 2 | 1 | 0 | 0 | 0 | 2
  Amylase increased | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 0
  Gamma-glutamyltransferase increased | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 1
  Hypercalcaemia | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
  Hypocalcaemia | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1
  Blood bilirubin increased | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
  Hyperkalaemia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1
  Lymphopenia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1
  Blood thyroid stimulating hormone increased | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  Hypoglycaemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Liver function test increased | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood phosphorus decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Febrile neutropenia | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Pancytopenia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  White blood cell count increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Blood creatine phosphokinase increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Hepatic enzyme increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypertransaminasaemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Leukopenia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Proteinuria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Blood albumin decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Blood iron decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Blood lactate dehydrogenase decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  International normalised ratio increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Megakaryocytes abnormal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Normocytic anaemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prothrombin time prolonged | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hypothyroidism | 0 | 0 | 1 | 2 | 2 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 2 | 1 | 0 | 2 | 0 | 1
  Hepatic cytolysis | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Blood lactate dehydrogenase increased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
  Pollakiuria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Blood urea increased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Haematuria | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Renal failure | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperthyroidism | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Myocardial infarction | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Adrenal insufficiency | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine renal clearance decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophil count increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Haemoglobin decreased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatraemia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Lymphadenopathy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Neutrophil count increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pancreatitis | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet count increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Troponin increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Type 1 diabetes mellitus | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vitamin B12 deficiency | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Azotaemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin conjugated increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood calcium decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Blood calcium increased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood chloride decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood chloride increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Blood fibrinogen decreased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood fibrinogen increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood glucose increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Blood magnesium decreased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood phosphorus increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Blood sodium decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Blood thrombin increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Brain natriuretic peptide increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Coagulation time prolonged | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Coagulopathy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Cushingoid | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Febrile bone marrow aplasia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Folate deficiency | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Haematocrit increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Haptoglobin increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hepatocellular injury | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hydronephrosis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hypercholesterolaemia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperlipasaemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypophysitis | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Iron deficiency | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pancreatitis acute | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Procalcitonin increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Protein total decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prothrombin time ratio increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Red blood cell count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Red blood cells urine positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Renal disorder | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Thyroiditis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Tri-iodothyronine increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Troponin T increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Type 2 diabetes mellitus | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs
Description: Number of participants with abnormal vital signs reported as TEAEs are reported. Abnormal vital signs are defined as any abnormal finding in the vital sign parameters (blood pressure, pulse rate, temperature, and respiration rate).
Time Frame: Day 1 thorugh 58.6 months (maximum observed duration)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg | Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg | Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg | Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg | Module 8 Cohort A.8.ATM: Ceralasertib 240 mg | Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg | Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 11 Cohort C.11.240: AZD6738 240 mg
Number analyzed (Participants) | 21 | 21 | 22 | 23 | 23 | 22 | 31 | 38 | 58 | 1 | 23 | 9 | 25 | 23 | 20 | 22 | 15 | 19 | 24 | 34 | 17 | 38
Participants
  Dyspnoea | 6 | 2 | 5 | 4 | 6 | 5 | 7 | 6 | 9 | 0 | 6 | 1 | 2 | 2 | 6 | 3 | 3 | 3 | 2 | 5 | 2 | 6
  Hypotension | 0 | 0 | 3 | 0 | 1 | 0 | 3 | 4 | 3 | 0 | 2 | 0 | 0 | 2 | 2 | 4 | 1 | 0 | 1 | 0 | 1 | 3
  Hypertension | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 5 | 1 | 0 | 0 | 0 | 0 | 0
  Tachycardia | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 4
  Dyspnoea exertional | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 0 | 1 | 1 | 0 | 1
  Blood pressure increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood pressure systolic increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bradycardia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Heart rate irregular | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypertensive crisis | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Abnormal Physical Examination Findings Reported as TEAEs
Description: Number of participants with abnormal physical examination findings reported as TEAEs are reported. Any new or aggravated clinically relevant abnormal medical finding at a physical examination as compared with the pre-dose assessment was reported as an AE.
Time Frame: Day 1 thorugh 58.6 months (maximum observed duration)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg | Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg | Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg | Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg | Module 8 Cohort A.8.ATM: Ceralasertib 240 mg | Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg | Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 11 Cohort C.11.240: AZD6738 240 mg
Number analyzed (Participants) | 21 | 21 | 22 | 23 | 23 | 22 | 31 | 38 | 58 | 1 | 23 | 9 | 25 | 23 | 20 | 22 | 15 | 19 | 24 | 34 | 17 | 38
Participants
  Weight decreased | 2 | 0 | 3 | 1 | 4 | 2 | 2 | 3 | 10 | 0 | 2 | 0 | 1 | 5 | 2 | 5 | 4 | 1 | 4 | 1 | 1 | 9
  Headache | 1 | 0 | 5 | 3 | 1 | 1 | 6 | 5 | 7 | 0 | 3 | 0 | 1 | 1 | 4 | 3 | 1 | 1 | 2 | 3 | 2 | 9
  Dizziness | 1 | 2 | 4 | 2 | 2 | 3 | 2 | 5 | 9 | 0 | 0 | 0 | 4 | 3 | 3 | 4 | 1 | 2 | 2 | 2 | 3 | 3
  Rash | 2 | 1 | 1 | 3 | 0 | 2 | 5 | 3 | 1 | 1 | 0 | 0 | 1 | 3 | 1 | 2 | 2 | 5 | 5 | 2 | 2 | 2
  Dry skin | 2 | 2 | 0 | 0 | 1 | 2 | 4 | 1 | 7 | 0 | 1 | 1 | 2 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 2 | 1
  Alopecia | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 4 | 7 | 0 | 1 | 0 | 1 | 2 | 0 | 1
  Dehydration | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 4 | 4 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1
  Hypoxia | 1 | 2 | 0 | 0 | 2 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  Myalgia | 2 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 3
  Rash maculo-papular | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Chronic obstructive pulmonary disease | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Tremor | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Erythema | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
  Rash pruritic | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Skin lesion | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Eczema | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Haematoma | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Skin hyperpigmentation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Psoriasis | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Skin exfoliation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Skin irritation | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Decubitus ulcer | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Orthostatic hypotension | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Skin disorder | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urticaria | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vena cava thrombosis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Breath sounds | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cardiac murmur | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Depressed level of consciousness | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dermatitis acneiform | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Dermatitis allergic | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dermatitis psoriasiform | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Ecchymosis | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphoedema | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nail disorder | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Peripheral ischaemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Petechiae | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Photosensitivity reaction | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Rash erythematous | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash macular | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Rash papular | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash pustular | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Seborrhoeic dermatitis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Skin discolouration | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Skin induration | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Skin mass | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Skin ulcer | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Superior vena cava syndrome | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Transient ischaemic attack | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

11. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Parameters Reported as TEAEs
Description: Number of participants with abnormal ECGs reported as TEAEs are reported.
Time Frame: Day 1 thorugh 58.6 months (maximum observed duration)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg | Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg | Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg | Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg | Module 8 Cohort A.8.ATM: Ceralasertib 240 mg | Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg | Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 11 Cohort C.11.240: AZD6738 240 mg
Number analyzed (Participants) | 21 | 21 | 22 | 23 | 23 | 22 | 31 | 38 | 58 | 1 | 23 | 9 | 25 | 23 | 20 | 22 | 15 | 19 | 24 | 34 | 17 | 38
Participants
  Sinus tachycardia | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 5
  Tachycardia | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 4
  Atrial fibrillation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
  Cardiac failure | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Electrocardiogram QT prolonged | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Cardiac arrest | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Arrhythmia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Ventricular extrasystoles | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Acute myocardial infarction | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Angina pectoris | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Atrial flutter | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Atrioventricular block second degree | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Bradycardia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Bundle branch block right | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Electrocardiogram RR interval prolonged | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Heart rate irregular | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myocardial ischaemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myocarditis | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myopericarditis | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supraventricular tachycardia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 through 61.55 months (maximum observed duration)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Arm/Group | Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg | Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg | Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg | Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg | Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg | Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg | Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg | Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg | Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg | Module 8 Cohort A.8.ATM: Ceralasertib 240 mg | Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg | Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg | Module 11 Cohort C.11.240: AZD6738 240 mg
All-Cause Mortality (participants affected / at risk) | 18/21 | 18/21 | 20/22 | 21/23 | 21/23 | 16/22 | 28/31 | 35/38 | 48/58 | 0/1 | 19/23 | 6/9 | 21/25 | 22/23 | 17/20 | 18/22 | 13/15 | 15/19 | 17/24 | 27/34 | 14/17 | 27/38
Serious Adverse Events (participants affected / at risk) | 10/21 | 7/21 | 8/22 | 7/23 | 12/23 | 8/22 | 11/31 | 11/38 | 17/58 | 0/1 | 7/23 | 1/9 | 6/25 | 10/23 | 10/20 | 7/22 | 7/15 | 7/19 | 13/24 | 12/34 | 1/17 | 17/38
Other Adverse Events (participants affected / at risk) | 19/21 | 19/21 | 19/22 | 21/23 | 22/23 | 19/22 | 30/31 | 34/38 | 55/58 | 1/1 | 19/23 | 5/9 | 22/25 | 23/23 | 20/20 | 20/22 | 15/15 | 17/19 | 24/24 | 30/34 | 16/17 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg (N=21) | Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg (N=21) | Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg (N=22) | Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg (N=23) | Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg (N=23) | Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg (N=22) | Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg (N=31) | Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg (N=38) | Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg (N=58) | Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg (N=1) | Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg (N=23) | Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg (N=9) | Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg (N=25) | Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg (N=23) | Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg (N=20) | Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg (N=22) | Module 8 Cohort A.8.ATM: Ceralasertib 240 mg (N=15) | Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg (N=19) | Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg (N=24) | Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg (N=34) | Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg (N=17) | Module 11 Cohort C.11.240: AZD6738 240 mg (N=38)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (3) | 2 (3) | 3 (3) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 6 (6)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Salmonellosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cor pulmonale (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal artery thrombosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myopericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Air embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Module 1 Cohort A.1.HRR: Durvalumab 1500 mg + Olaparib 300 mg (N=21) | Module 1 Cohort A.1.LKB: Durvalumab 1500 mg + Olaparib 300 mg (N=21) | Module 1 Cohort B.1.PRI: Durvalumab 1500 mg + Olaparib 300 mg (N=22) | Module 1 Cohort B.1.ACQ: Durvalumab 1500 mg + Olaparib 300 mg (N=23) | Module 2 Cohort B.2.PRI: Durvalumab 1500 mg + Danvatirsen 200 mg (N=23) | Module 2 Cohort B.2.ACQ: Durvalumab 1500 mg + Danvatirsen 200 mg (N=22) | Module 3 Cohort A.3.ATM: Durvalumab 1500 mg + AZD6738 240 mg (N=31) | Module 3 Cohort B.3.PRI: Durvalumab 1500 mg + AZD6738 240 mg (N=38) | Module 3 Cohort B.3.ACQ: Durvalumab 1500 mg + AZD6738 240 mg (N=58) | Module 4 Cohort A.4.RIC: Durvalumab 1500 mg + Vistusertib 125 mg (N=1) | Module 5 Cohort A.5.73H: Durvalumab 1500 mg + Oleclumab 3000 mg (N=23) | Module 5 Cohort B.5.PRI: Durvalumab 1500 mg + Oleclumab 3000 mg (N=9) | Module 5 Cohort B.5.ACQ: Durvalumab 1500 mg + Oleclumab 3000 mg (N=25) | Module 6 Cohort A.6.HER2e: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg (N=23) | Module 6 Cohort A.6.HER2m: Durvalumab 1120 mg + Trastuzumab Deruxtecan 5.4mg/kg (N=20) | Module 7 Cohort B.7.ACQ: Durvalumab 1500 mg + Cediranib 20 mg (N=22) | Module 8 Cohort A.8.ATM: Ceralasertib 240 mg (N=15) | Module 9 Cohort B.9.PRI: Durvalumab 1500 mg + Ceralasertib 240 mg (N=19) | Module 9 Cohort B.9.ACQ: Durvalumab 1500 mg + Ceralasertib 240 mg (N=24) | Module 10 Cohort C.10.160: Durvalumab 1500 mg + Ceralasertib 160 mg (N=34) | Module 10 Cohort C.10.240: Durvalumab 1500 mg + Ceralasertib 240 mg (N=17) | Module 11 Cohort C.11.240: AZD6738 240 mg (N=38)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 2 (2) | 2 (2) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 6 (6) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 5 (5) | 9 (12) | 1 (1) | 2 (2) | 2 (2)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (5) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (6) | 3 (4)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 1 (2) | 1 (1) | 0 (0) | 4 (7) | 0 (0) | 2 (8) | 2 (3)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (4) | 1 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 1 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 2 (3) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 2 (2)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (6)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (5) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Megakaryocytes abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 0 (0) | 2 (2) | 1 (2) | 2 (5) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 4 (8) | 1 (3) | 5 (11) | 0 (0) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 2 (2) | 2 (2) | 3 (3) | 10 (12) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 2 (2) | 5 (6) | 4 (4) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 9 (10)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 4 (4) | 3 (3) | 8 (8) | 4 (4) | 3 (4) | 6 (6) | 10 (10) | 22 (24) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 10 (12) | 7 (8) | 5 (6) | 7 (7) | 4 (4) | 7 (8) | 6 (6) | 5 (7) | 15 (17)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 2 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 3 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 5 (7) | 1 (2) | 2 (2) | 1 (1) | 2 (5) | 3 (3) | 1 (1) | 4 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (4) | 3 (3) | 0 (0) | 3 (4) | 2 (2) | 8 (11) | 3 (3) | 4 (6) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (4) | 2 (2) | 4 (4) | 1 (1) | 8 (9) | 3 (3) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 3 (4) | 5 (5) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 2 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 7 (11) | 7 (12) | 5 (5) | 7 (10) | 4 (4) | 4 (5) | 10 (11) | 9 (10) | 19 (22) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 7 (9) | 12 (20) | 1 (1) | 12 (16) | 8 (9) | 12 (14) | 5 (6) | 7 (7) | 15 (21)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 5 (5) | 9 (11) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 3 (3) | 4 (4) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 5 (5) | 3 (3) | 1 (1) | 1 (1) | 6 (6) | 5 (5) | 7 (9) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 3 (7) | 2 (2) | 9 (11)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypotonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Neuropsychological symptoms (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (6) | 2 (2) | 4 (4) | 4 (4) | 8 (10) | 3 (3) | 6 (6) | 9 (9) | 0 (0) | 4 (4) | 1 (1) | 2 (3) | 4 (4) | 2 (2) | 3 (3) | 1 (1) | 3 (4) | 2 (2) | 3 (3) | 1 (1) | 5 (8)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 3 (3) | 4 (5) | 4 (4) | 5 (5) | 6 (6) | 6 (7) | 6 (6) | 0 (0) | 6 (6) | 1 (1) | 2 (2) | 2 (2) | 5 (5) | 3 (3) | 3 (3) | 3 (3) | 2 (3) | 3 (3) | 2 (2) | 6 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 4 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 5 (6) | 1 (1) | 6 (7) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 7 (7) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (5) | 1 (1) | 7 (7) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 5 (5) | 3 (3) | 4 (5) | 2 (2) | 4 (4) | 0 (0) | 4 (5) | 0 (0) | 6 (7) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 6 (7) | 4 (5) | 2 (2) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (3) | 3 (3) | 0 (0) | 2 (2) | 5 (8) | 3 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (4) | 2 (5) | 5 (5) | 5 (5) | 2 (2) | 2 (2) | 2 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 3 (3) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (7) | 3 (3) | 5 (6) | 3 (3) | 2 (2) | 2 (3) | 6 (6) | 5 (5) | 16 (16) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 5 (7) | 2 (2) | 0 (0) | 3 (3) | 1 (2) | 1 (2) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 2 (3) | 4 (6) | 5 (7) | 5 (7) | 3 (3) | 8 (13) | 9 (11) | 11 (22) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 8 (10) | 5 (6) | 8 (13) | 1 (1) | 3 (4) | 7 (7) | 6 (8) | 3 (3) | 8 (15)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 4 (4)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (13) | 7 (8) | 10 (14) | 16 (18) | 2 (2) | 1 (1) | 19 (42) | 19 (25) | 34 (40) | 0 (0) | 4 (4) | 0 (0) | 4 (4) | 18 (28) | 12 (17) | 4 (5) | 10 (11) | 5 (6) | 10 (14) | 14 (24) | 6 (10) | 22 (33)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (12) | 4 (6) | 7 (12) | 8 (11) | 1 (1) | 2 (2) | 10 (12) | 11 (13) | 15 (28) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 8 (18) | 9 (13) | 1 (2) | 4 (4) | 5 (6) | 6 (8) | 9 (13) | 5 (6) | 12 (18)
Asthenia (General disorders) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 7 (8) | 6 (6) | 11 (11) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 4 (4) | 5 (5) | 4 (4) | 5 (6) | 1 (1) | 10 (10)
Catheter site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Fatigue (General disorders) | 10 (10) | 5 (5) | 5 (5) | 9 (11) | 3 (3) | 6 (8) | 8 (10) | 6 (7) | 16 (37) | 0 (0) | 2 (2) | 3 (3) | 8 (9) | 8 (11) | 9 (11) | 10 (12) | 6 (7) | 4 (4) | 9 (9) | 2 (2) | 3 (3) | 16 (22)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 2 (2) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 2 (3) | 4 (6) | 3 (3) | 5 (5) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 8 (12)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contrast media reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (5) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal foot infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Module 4 was prematurely discontinued by the sponsor for strategic reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript; it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT03334617/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT03334617/SAP_001.pdf